CLINICAL TRIAL: NCT02744352
Title: Comparison Between Single Shot Versus Continuous Infraclavicular Brachial Plexus Block for Postoperative Analgesia After Distal Radius Fracture: A Prospective Randomized Open Label Study
Brief Title: Single Shot vs Catheter Infraclavicular Brachial Plexus Block After Distal Radius Fracture Repair
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: prior to its planned completion as anticipated by the protocol due to lack of resources
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 823323
Record Dates: First submitted 2016-03-23; First posted 2016-04-20 (Estimated); Results first posted 2020-03-25 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Distal Radius Fracture; Post Operative Pain Control
Keywords: infraclavicular brachial plexus block; quality of recovery score; pain score; disability assessment of shoulder and hand questionnaire
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- continuous IBP block (Active Comparator): Subjects will receive 60 hour continuous infraclavicular brachial plexus block (0.2% of ropivacaine at 8 milliliter/hour) with initial four intermittent 5ml bolus (20ml) of 0.5% Ropivicaine given preoperatively to help with operative and postoperative pain
  Interventions: Drug: 20ml bolus of 0.5% ropivicaine; Drug: 0.2% of ropivacaine at 8 milliliter/hour
- single shot IBP block (Active Comparator): Subjects will receive single shot infraclavicular brachial plexus block with 20ml bolus of 0.5% ropivicaine given preoperatively to help with operative and postoperative pain
  Interventions: Drug: 20ml bolus of 0.5% ropivicaine

INTERVENTIONS:
Drug: 20ml bolus of 0.5% ropivicaine — Local anesthetic
Drug: 0.2% of ropivacaine at 8 milliliter/hour — Local anesthetic
  Arms: continuous IBP block

SUMMARY:
The purpose of this study is to compare infraclavicular brachial plexus shot single shot block to continuous catheter nerve block done in adult patients who have under gone surgery to repair distal radius fractures. Visual analogue scores, opioid consumption, quality of recovery and quality of sleep up to 72 hours post operatively will be used for comparison.

DETAILED DESCRIPTION:
If the patient is willing to participate and signs the consent, he/she will be randomized to one of the two treatment groups:

1. Single shot block
2. Continuous catheter

In the institution investigators usually advocate for regional anesthesia and intravenous sedation for the repair of open fracture of the distal radius.

Patients will be monitored during block performance with standard ASA monitors. All patients will receive 2 L of oxygen via a nasal cannula. Sedatives will be titrated to effect. Midazolam 1-2 mg, and fentanyl 50-100 mcg will be used for sedation.

Block time out will be preformed according to standard operating procedure. All blocks will be done under ultrasound guidance. Sonosite S nerve machine will be used with a low frequency curvilinear (C5) US probe with 2-5 MHZ frequency. Both single shot and continuous ICB will be performed according to the SOP in the department. Ultrasound survey of the deltopectoral groove below the clavicle will take place. The axillary artery and the three cords (posterior, medial and lateral) of the brachial plexus will be identified in short axis view deeper to the pectoralis minor muscle.

For single shot blocks: A 4 inch 21 gauge single shot (B-Braun) needle will be introduced in-plane towards the posterior cord of the brachial plexus and 1-2 mL of dextrose 5% (D5%) bolus will be used to verify correct placement of the needle in the vicinity of the posterior cord and adequate spread pattern to both lateral and medical cord. 20 ml of of Ropivicaine 0.5% will be injected through the needle with intermittent aspiration after each 5 ml bolus injection.

For the continuous block: A 4 gauge 18 inch tuohy needle ( B -Braun) will be introduced towards the posterior cord as above. When the needle tip and the pattern of spread is confirmed using D5% solution, a 21 gauge catheter will be introduced 2 cm beyond the needle tip under ultrasound visualization. The needle will be withdrawn over the catheter. Injection of a total of 20 ml of ropivacaine 0.5% ( in divided 5 ml boluses with intermittent aspiration) will take place through the catheter while observing the spread of local anesthetic under ultrasound. The catheter hub will be affixed to the upper lateral chest with sterile occlusive dressings and an anchoring device.

Block success will be defined as a change in cutaneous sensation to touch with an alcohol pad in the posterior, medial and lateral cord distribution over the forearm and the hand within 30min after injection. Subjects with successful catheter placement per protocol and nerve block onset will be retained in the study. Subjects with a failed catheter insertion or misplaced catheter indicated by a lack of sensory changes will have their catheter replaced or will be single shot blocked and withdrawn from the study.

Intraoperative sedation will consist of intermittent boluses of midazolam (1-2 mg), fentanyl (50-100 mcg) and propofol infusion, titrates to sedation and patient comfort (25-50 mcg/kg/min).

All patients will receive prophylaxis for postoperative nausea and vomiting (PONV) during surgery. The protocol for prophylaxis against PONV includes administration of 4 mg of dexamethasone after induction of anesthesia and 4 mg of ondansetron 20 minutes before recovery from anesthesia. Dexamethasone is withheld if the patient has poorly controlled diabetes mellitus (DM). Uncontrolled DM will be defined as random blood glucose above 250 mg/dl.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for open reduction and internal fixation of a distal radius fracture
* American Society of Anesthesiologists (ASA) physical status I -III
* Mentally competent and able to give consent for enrollment in the study

Exclusion Criteria:

* Patient younger than 18 years old
* Allergy to local anesthetics, systemic opioids (fentanyl, morphine, hydromorphone and any of the drugs included in the standard of care
* Patients opting to go under general anesthesia and those refusing the block
* Chronic pain syndromes; Patients will be defined to have chronic pain if they are using regular daily doses of systemic narcotics for the past 6 months prior to the surgery
* BMI of 40 or more

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-10-05 (Actual); Study Completion 2018-10-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nabil M Elkassabany, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Continuous IBP Block | Single Shot IBP Block
Started | 4 | 4
Completed | 4 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Continuous IBP Block | Single Shot IBP Block | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 4 | 8
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 2 | 1 | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 4

OUTCOME MEASURES:

1. Primary Outcome: Pain Scores as Measured by the Visual Analog Scale
Description: Pain scores at rest and with movement.
Time Frame: 72 hours
Population: Analysis not done because study terminated prior to treatment.
Arm/Group | Continuous IBP Block | Single Shot IBP Block
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Participants Need for Pain Relief as Measured by Opiate Consumption
Description: Amount of opiate consumption
Time Frame: 72 hours
Population: Analysis not done because study terminated prior to treatment.
Arm/Group | Continuous IBP Block | Single Shot IBP Block
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Quality of Recovery Score
Description: Score of QoR survey to determine recovery status
Time Frame: 72 hours
Population: Study was terminated before patient analysis and follow ups were completed.
Arm/Group | Continuous IBP Block | Single Shot IBP Block
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Number of Subjects With Insomnia as Measured by Sleep Questionnaire
Description: Quality of sleep first 2 nights post surgery
Time Frame: 48 hours
Population: Analysis not done because study terminated prior to treatment.
Arm/Group | Continuous IBP Block | Single Shot IBP Block
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Range of Motion as Measured by the Disability Assessment of Shoulder and Hand Questionnaire
Description: Dash questionnaire to measure range of motion of the wrist and fingers 3 months after surgery
Time Frame: 3 months
Population: Analysis not done because study terminated prior to treatment.
Arm/Group | Continuous IBP Block | Single Shot IBP Block
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 2 Years
Arm/Group | Continuous IBP Block | Single Shot IBP Block
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 0/4 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-05-29): https://cdn.clinicaltrials.gov/large-docs/52/NCT02744352/Prot_SAP_000.pdf
  • Informed Consent Form (2017-08-24): https://cdn.clinicaltrials.gov/large-docs/52/NCT02744352/ICF_001.pdf